CLINICAL TRIAL: NCT03735420
Title: Xanthohumol Metabolism and Signature (XMaS) in Healthy Adults
Brief Title: Xanthohumol Metabolism and Signature
Acronym: XMaS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Oregon State University (Other); Pacific Northwest National Laboratory (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ryan Bradley, Director, Helfgott Research Institute, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RB9718
Record Dates: First submitted 2018-10-11; First posted 2018-11-08 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: xanthohumol; gut microbiome; inflammation
MeSH Terms: conditions — Inflammation | interventions — xanthohumol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either encapsulated xanthohumol in a rice protein vehicle, or an identical capsule containing vehicle alone.
Who Masked: Participant, Investigator
Masking Description: Randomization will occur in up to 8 blocks of 4 based on biological sex. Initial randomization series will be generated using readily available random sequence generators designed to do so. A series of sequential envelopes will be generated, each containing the allocation for one participant. Envelopes will be opaque and signed across the seal. The randomization "code" will be kept in a sealed envelope with a signature across the label and dated the day of creation. Study product and comparator (placebo) will be compounded and placed in identical opaque capsules outside the institution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xanthohumol (Experimental): Participants will receive 24 mg of 98% pure xanthohumol in a rice protein vehicle by mouth once daily with the first daily meal.
  Interventions: Drug: Xanthohumol
- Placebo oral capsule (Placebo Comparator): Participants will receive vehicle (rice protein) by mouth once daily with the first daily meal.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Xanthohumol — The xanthohumol supplement will be administered in a capsule. Participants in the experimental arm will consume the capsule once per day, with the first meal. The intervention will extend for 8 weeks.
  Arms: Xanthohumol
Drug: Placebo oral capsule — The placebo (vehicle) will be administered in a capsule. Participants in the placebo arm will consume the capsule once per day, with the first meal.
  Other Names: Vehicle
  Arms: Placebo oral capsule

SUMMARY:
A pilot study to assess the safety and tolerability of oral xanthohumol in humans, to identify a biological signature of xanthohumol exposure, and to characterize the role of xanthohumol metabolism by intestinal microorganisms in that signature.

DETAILED DESCRIPTION:
This is a double-masked, placebo controlled, randomized clinical trial of xanthohumol, which is a constituent of hops (Humulus lupulus). Hops and its constituents have a long history of use for a variety of conditions. However, knowledge is limited regarding the measurable biological markers of human exposure, and the role of xanthohumol metabolism by microorganisms present in the gut. This information is necessary for the development of xanthohumol as a potential therapeutic intervention in conditions such as inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged 21-50 years
* Willing to take isolated xanthohumol as a dietary supplement for 8 weeks
* Willing to have blood drawn semi-weekly and to fast for 10-12 hours before blood draws
* Willing and able to collect semi-weekly stool samples at home
* Able to speak, read, and understand English
* Must be able to provide written informed consent
* Non-smokers (including tobacco and Cannabis products, combusted or vaporized)

Exclusion Criteria:

* History of any chronic disease including, but not limited to: diabetes (type 1 or 2); uncontrolled hypertension; coronary artery disease resulting in angina; cardiovascular disease requiring percutaneous coronary intervention (PCI), bypass, or past myocardial infarction or stroke; blood disease including current anemia; cancer (except non-melanoma skin cancer) within the last year or still requiring chemotherapy or hormonal therapy; chronic kidney disease; liver disease including viral hepatitis, non-alcoholic fatty liver disease, or alcoholic hepatitis/cirrhosis; any immunocompromising condition including human immunodeficiency virus/acquired immunodeficiency syndrome or organ transplant requiring anti-rejection medications; chronic osteoarthritis requiring joint replacement or daily use of NSAIDs; chronic endocrine condition including but not limited to: Cushing's, Addison's, Hashimoto's thyroiditis, Grave's disease, etc.
* Body Mass Index (BMI) less than 20 (underweight) or greater than 30 (obese)
* Consumption of more than 1 microbrew beer per day
* Use of NSAIDs more than once per week for headaches, routine aches/pains, etc.
* Use of any prescription drugs, including oral contraceptives (due to potential interference with mechanisms under investigation)
* Use of prescription opioids for any reason within the past 3 months
* Use of prescription corticosteroids for any reason within the past 3 months
* Free of acute viral or bacterial infection, or recent infection within the last 14 days or still requiring prescription medication for treatment
* Free of recent acute trauma occurring within the last 14 days
* Currently or recently (within last 14 days) taking any dietary supplements containing xanthohumol flavonoids, or other known herbal "anti-inflammatories" including: curcumin, turmeric, fenugreek, hops, rosemary, ginger, white willow, Devil's claw, fish oil (doses>1 g/day), or quercetin. Candidates will be given the option to "wash out" for 14 days and re-contact the study team.
* Currently receiving intravenous nutrition support therapy (or within the last 30 days)
* Currently taking anti-coagulant or anti-platelet prescription medications (or they were taken within the last 30 days)
* Currently taking antibiotic, antiparasitic, or antifungal medications orally or intravenously (or they were taken within the last 30 days)
* Initiation of or changes to supplements or medications within 30 days prior to screening
* Initiation of or changes to an exercise regimen within 30 days prior to screening
* Initiation of or changes to a food plan within 30 days prior to screening
* Current involvement or within 30 days prior to screening of a significant diet or weight loss program, such as NutriSystem, Jenny Craig, Atkin's or other low-carb diet programs, or very low-calorie liquid diet programs (such as optifast, medifast, and/or HMR)
* Hospitalization (for any reason other than an elective medical procedure) within 3 months prior to screening
* Gastrointestinal surgery within 3 months prior to screening
* Undergoing UV therapy (e.g. treatment for skin conditions such as psoriasis).
* Engaging in vigorous exercise more than 6 hours per week.
* Women who are lactating, pregnant or planning pregnancy within the next four months
* Typical intake of more than 2 alcohol-containing beverages per day, more than 14 per week, or more than 4 in any single day within the past 28 days
* Use of recreational drugs/substances (such as but not limited to cocaine, phencyclidine (PCP), and methamphetamine) within 30 days of screening
* Currently participating in another interventional research study or participated in another interventional study within 30 days of screening

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2024-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, MPH, Principal Investigator — National University of Natural Medicine
Locations (1):
- Helfgott Research Institute National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We will use the University of California San Diego (UCSD) Metabolomics Workbench for sharing metabolomics datasets and results (including raw data matrices, platform information, and associated metadata).
  For activity-based proteomics data, we will use PRIDE or the MassIVE data repository at UCSD.
  Nucleic acid sequence data will be submitted to the National Center for Biotechnology Information (NCBI) Short Read Archive.
  Gene expression data will be submitted to Gene expression Omnibus at NCBI. Microbiome metadata will be deposited into database of Genotypes and Phenotypes.
  Metagenomic nucleic acid sequence data will additionally be deposited in Metagenomic Rapid Annotations using Subsystems Technology (MG-RAST) at Argonne National Laboratory, along with associated metadata.
  Microbiome summary files (e.g., tables cataloging: sample metadata, taxon or protein family abundances across samples) publicly available through github.
Time Frame: We will share our data no later than on acceptance of the first publication of the findings from the respective data set(s).
Access Criteria: All indicated repositories are freely available to the research community.

REFERENCES:
- [Derived] Jamieson PE, Smart EB, Bouranis JA, Choi J, Danczak RE, Wong CP, Paraiso IL, Maier CS, Ho E, Sharpton TJ, Metz TO, Bradley R, Stevens JF. Gut enterotype-dependent modulation of gut microbiota and their metabolism in response to xanthohumol supplementation in healthy adults. Gut Microbes. 2024 Jan-Dec;16(1):2315633. doi: 10.1080/19490976.2024.2315633. Epub 2024 Feb 15. PMID 38358253
- [Derived] Bradley R, Langley BO, Ryan JJ, Phipps J, Hanes DA, Stack E, Jansson JK, Metz TO, Stevens JF. Xanthohumol microbiome and signature in healthy adults (the XMaS trial): a phase I triple-masked, placebo-controlled clinical trial. Trials. 2020 Oct 7;21(1):835. doi: 10.1186/s13063-020-04769-2. PMID 33028396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xanthohumol | Placebo Oral Capsule
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xanthohumol | Placebo Oral Capsule | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.06 (6.45) | 33.14 (5.36) | 30.97 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 12 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Body mass index [Mean (Standard Deviation); unit: kilogram per meters-squared (kg/m2)] | 23.41 (2.23) | 23.30 (2.57) | 23.36 (2.36)
Heart rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 64.50 (11.78) | 61.07 (8.30) | 62.90 (10.28)
Weight [Mean (Standard Deviation); unit: kilograms] | 69.82 (10.33) | 70.60 (14.59) | 70.18 (12.28)
Height [Mean (Standard Deviation); unit: meters] | 1.73 (0.12) | 1.73 (0.11) | 1.73 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Inflammatory Markers
Description: Circulating pro-inflammatory cytokine concentrations (tumor necrosis factor (TNF)-α, interleukin (IL)-1 beta, IL-6, IL-8, IL-10, and IL-12p70), will be measured simultaneously with a flow cytometry-based multiplex assay. The measures were assessed at Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks; weeks 2, 4, 6, and 8 reported
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
picogram per milliliter (pg/mL)
  Week 2: Interleukin 1-beta (IL-1b) | 220 (358) | -2463 (12960)
  Week 4: IL-1b | 172 (677) | -3153 (12490)
  Week 6: IL-1b | 2368 (7689) | -620 (16359)
  Week 8: IL-1b | -133 (328) | -3624 (12306)
  Week 2: Interleukin 6 (IL-6) | -54 (252) | -784 (2795)
  Week 4: IL-6 | -79 (263) | -684 (2552)
  Week 6: IL-6 | -51 (251) | -764 (2802)
  Week 8: IL-6 | 3565 (12594) | -784 (2792)
  Week 2: Interleukin 8 (IL-8) | 1796 (6380) | -5914 (22847)
  Week 4: IL-8 | -7 (352) | 7669 (62489)
  Week 6: IL-8 | 276 (840) | -6955 (25976)
  Week 8: IL-8 | 2639 (6116) | -6882 (25878)
  Week 2: Interleukin 10 (IL-10) | 76 (273) | -46 (180)
  Week 4: IL-10 | 10 (44) | -34 (150)
  Week 6: IL-10 | -2 (17) | -49 (177)
  Week 8: IL-10 | -3 (13) | -43 (171)
  Week 2: Interleukin 12p70 (IL-12p70) | 2 (9) | 25 (154)
  Week 4: IL-12p70 | 3 (12) | -7 (52)
  Week 6: IL-12p70 | -2 (12) | -14 (46)
  Week 8: IL-12p70 | 1 (9) | 0 (55)
  Week 2: Tumor Necrosis Factor Alpha (TNFa) | 2 (9) | -8 (124)
  Week 4: TNFa | -3 (9) | -28 (100)
  Week 6: TNFa | -4 (10) | -23 (102)
  Week 8: TNFa | -1 (8) | -25 (100)

2. Primary Outcome: Incidence of Intervention-attributable Adverse Events [Safety and Tolerability]
Description: Self-reported adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events. Reported as: New onset "FDA serious" adverse events (Grade 1); New onset "moderate" adverse events (Grade 2). The measures were assessed at Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks; weeks 2, 4, 6, and 8 reported.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Number; unit: Adverse events
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
Adverse events
  Week 2 Grade 1 | 12 | 9
  Week 2 Grade 2 | 2 | 2
  Week 4 Grade 1 | 18 | 9
  Week 4 Grade 2 | 0 | 3
  Week 6 Grade 1 | 18 | 11
  Week 6 Grade 2 | 8 | 2
  Week 8 Grade 1 | 5 | 0
  Week 8 Grade 2 | 2 | 2

3. Secondary Outcome: Change in Levels of Metabolic Byproducts of Xanthohumol: Plasma and Urine
Description: Xanthohumol and xanthohumol metabolites in blood, urine and stool, will be measured by ultra-high performance liquid chromatography-quadrupole time-of-flight mass spectrometry. Metabolites include 6-prenylnaringenin (6-PN), 8-prenylnaringenin (8-PN), dihydroxanthohumol (DXN), desmethyldihydroxanthohumol (DDXN), isoxanthohumol (IXN), and xanthohumol (XN). The measures were assessed at Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks; baseline, weeks 2, 4, 6, and 8 reported for urine and plasma.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: nanograms per millileter (ng/mL)
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
nanograms per millileter (ng/mL)
  Urinary 6-Prenylnaringenin (6-PN): Baseline | 0 (0) | 0 (0)
  Urinary 6-PN: Week 2 | 0 (0) | 0 (0)
  Urinary 6-PN: Week 4 | .591 (2.132) | 0 (0)
  Urinary 6-PN: Week 6 | 0 (0) | 0 (0)
  Urinary 6-PN: Week 8 | 0 (0) | 0 (0)
  Urinary 8-Prenylnaringenin (8-PN): Baseline | 0 (0) | 0 (0)
  Urinary 8-PN: Week 2 | 6.811 (12.029) | 1.412 (3.877)
  Urinary 8-PN: Week 4 | 6.588 (0.840) | 0 (0)
  Urinary 8-PN: Week 6 | 7.196 (14.662) | 0 (0)
  Urinary 8- PN Week 8 | 4.725 (7.769) | 0 (0)
  Urinary Dihydroxanthohumol (DXN): Baseline | 0 (0) | .086 (.312)
  Urinary DXN: Week 2 | .562 (.542) | 0 (0)
  Urinary DXN: Week 4 | .561 (.522) | 0 (0)
  Urinary DXN: Week 6 | .410 (.325) | 0 (0)
  Urinary DXN: Week 8 | 2.043 (4.702) | .016 (.059)
  Urinary Desmethyldihydroxanthohumol (DDXN): Baseline | .042 (.152) | 0 (0)
  Urinary DDXN: Week 2 | .041 (.148) | 0 (0)
  Urinary DDXN: Week 4 | .036 (.131) | 0 (0)
  Urinary DDXN: Week 6 | 0 (0) | 0 (0)
  Urinary DDXN: Week 8 | .071 (.257) | .023 (.083)
  Urinary Isoxanthohumol (IXN): Baseline | 2.237 (4.364) | .299 (1.080)
  Urinary IXN: Week 2 | 94.120 (82.500) | 2.121 (4.001)
  Urinary IXN: Week 4 | 103.920 (75.201) | .494 (1.782)
  Urinary IXN: Week 6 | 66.628 (41.899) | .281 (1.012)
  Urinary IXN: Week 8 | 95.756 (83.275) | .484 (1.745)
  Urinary Xanthohumol (XN) Baseline | 1.952 (13.967) | 0 (0)
  Urinary XN: Week 2 | 21.280 (12.112) | 4.666 (16.440)
  Urinary XN: Week 4 | 14.908 (8.667) | .124 (.448)
  Urinary XN: Week 6 | 19.979 (12.242) | 0 (0)
  Urinary XN: Week 8 | 19.952 (13.967) | 0 (0)
  Plasma 6-Prenylnaringenin (6PN): Baseline | 0 (0) | 0 (0)
  Plasma 6-PN: Week 2 | 0 (0) | 0 (0)
  Plasma 6-PN: Week 4 | 0 (0) | 0 (0)
  Plasma 6-PN: Week 6 | 0 (0) | 0 (0)
  Plasma 6-PN: Week 8 | 0 (0) | 0 (0)
  Plasma 8-Prenylnaringenin: Baseline | 1.302 (3.034) | 0 (0)
  Plasma 8-PN: Week 2 | 1.503 (3.340) | 0 (0)
  Plasma 8-PN: Week 4 | .840 (3.144) | 0 (0)
  Plasma 8-PN: Week 6 | 1.001 (2.563) | 0 (0)
  Plasma 8-PN: Week 8 | 1.302 (3.034) | 0 (0)
  Plasma Dihydroxanthohumol (DXN): Baseline | 0 (0) | 0 (0)
  Plasma DXN: Week 2 | .968 (3.622) | 0 (0)
  Plasma DXN: Week 4 | 0 (0) | 0 (0)
  Plasma DXN: Week 6 | 0 (0) | 7.288 (25.245)
  Plasma DXN: Week 8 | 0 (0) | 0 (0)
  Plasma Desmethyldihydroxanthohumol (DDXN): Baseline | 0 (0) | 0 (0)
  Plasma DDXN: Week 2 | 0 (0) | 0 (0)
  Plasma DDXN: Week 4 | 0 (0) | 0 (0)
  Plasma DDXN: Week 6 | 0 (0) | 0 (0)
  Plasma DDXN: Week 8 | 0 (0) | 0 (0)
  Plasma Isoxanthohumol (IXN): Baseline | 0 (0) | .275 (.992)
  Plasma IXN: Week 2 | 7.864 (4.135) | 0 (0)
  Plasma IXN: Week 4 | 6.999 (3.514) | 0 (0)
  Plasma IXN: Week 6 | 6.140 (3.565) | 0 (0)
  Plasma IXN: Week 8 | 8.174 (3.794) | 0 (0)
  Plasma Xanthohumol (XN): Baseline | 0 (0) | .365 (.974)
  Plasma XN: Week 2 | 7.156 (3.888) | 1.325 (3.424)
  Plasma XN: Week 4 | 6.784 (3.497) | 0 (0)
  Plasma XN: Week 6 | 5.810 (3.153) | .822 (2.304)
  Plasma XN: Week 8 | 5.796 (3.188) | 0 (0)

4. Secondary Outcome: Change in Levels of Metabolic Byproducts of Xanthohumol: Stool
Description: Xanthohumol and xanthohumol metabolites in blood, urine and stool, will be measured by ultra-high performance liquid chromatography-quadrupole time-of-flight mass spectrometry. Metabolites include 6-prenylnaringenin (6-PN), 8-prenylnaringenin (8-PN), dihydroxanthohumol (DXN), desmethyldihydroxanthohumol (DDXN), isoxanthohumol (IXN), and xanthohumol (XN). The measures were assessed at Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks; baseline, weeks 2, 4, 6, and 8 reported for urine and plasma. As stool metabolites have not yet been analyzed, data will be released upon assessment.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Reporting Status: Not Posted, anticipated posting 2024-12

5. Secondary Outcome: Bile Acids
Description: Bile acid concentrations in blood and feces, will be measured by ultra-high performance liquid chromatography-quadrupole time-of-flight mass spectrometry, and expressed as mean change over time from baseline.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Reporting Status: Not Posted, anticipated posting 2024-12

6. Secondary Outcome: Gut Inflammation
Description: Fecal calprotectin, a protein associated with gut inflammation and irritable gut syndrome, will be measured by enzyme-linked immunosorbent assay, and expressed as mean change over time from baseline.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: microgram per milligram (ug/mg)
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
microgram per milligram (ug/mg)
  Baseline | 12.8 (2.7) | 35.2 (76.7)
  Week 2 | 12.4 (1.5) | 19.9 (21.8)
  Week 4 | 13.4 (3.9) | 12.7 (2.5)
  Week 6 | 12.7 (2.5) | 14.3 (5.4)
  Week 8 | 15.2 (10.3) | 13.2 (2.6)

7. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: Aspartate aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. Reported as mean change from baseline.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mgdL)
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
milligrams per deciliter (mgdL)
  Week 2 | 22.9 (13.5) | 15.4 (2.6)
  Week 4 | 18.3 (5.1) | 15.3 (3.01)
  Week 6 | 21.1 (8.9) | 16.4 (3.2)
  Week 8 | 18.4 (5.8) | 15.5 (2.6)

8. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: Alanine aminotransferase is an enzyme that is often measured in blood as an indication of liver toxicity. Reported as mean change from baseline.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: milligrams per decileter (mg/dL)
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
milligrams per decileter (mg/dL)
  Week 2 | 18.0 (15.1) | 14.9 (3.8)
  Week 4 | 16.1 (7.5) | 14.0 (3.81)
  Week 6 | 16.4 (7.5) | 15.4 (5.11)
  Week 8 | 15.1 (9.2) | 12.9 (2.84)

9. Secondary Outcome: Gamma-Glutamyl Transferase (GGT)
Description: Gamma-glutamyl transferase is an enzyme that is often measured in blood as an indication of liver toxicity. Reported as mean change from baseline.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
Measure: Mean (Standard Deviation); unit: milligrams per decileter (mg/dL)
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
milligrams per decileter (mg/dL)
  Week 2 | 12.1 (3.40) | 11.8 (4.58)
  Week 4 | 12.3 (4.30) | 11.8 (5.82)
  Week 6 | 12.9 (4.74) | 12.3 (6.92)
  Week 8 | 12.1 (4.52) | 11.8 (5.00)

10. Secondary Outcome: Estimated Glomerular Filtration Rate
Description: Glomerular filtration rate is estimated based on blood creatinine concentration per standard nephrology practice. Reported as mean change from baseline.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks
Measure: Mean (Standard Deviation); unit: millileters per minute (mL/min)
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
millileters per minute (mL/min)
  Week 2 | 108.7 (11.3) | 112.0 (12.9)
  Week 4 | 110.6 (11.4) | 111.8 (12.1)
  Week 6 | 109.2 (10.2) | 111.4 (11.2)
  Week 8 | 108.4 (11.9) | 111.8 (13.8)

11. Secondary Outcome: Blood Urea Nitrogen to Creatinine Ratio
Description: Blood urea nitrogen (BUN) : creatinine (Cr) is a ratio of serum concentrations of two compounds associated with renal function. Reported as mean change from baseline.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: Ratio of BUN (mg/dL) to Cr (mg/dL)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
Ratio of BUN (mg/dL) to Cr (mg/dL)
  Baseline | 15.6 (40.8) | 14.5 (25.2)
  Week 2 | 16.4 (29.0) | 15.5 (32.4)
  Week 4 | 15.2 (31.5) | 15.3 (26.4)
  Week 6 | 14.8 (41.4) | 14.5 (23.4)
  Closeout | 14.5 (30.9) | 14.7 (26.3)

12. Secondary Outcome: Complete Blood Count Abnormals
Description: Enumeration of the various subtypes of blood cells (i.e., red blood cells, white blood cells, and platelets), plus indices including mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), and hematocrit. Reported as: % abnormal (i.e., number of participants with an abnormal value compared to the number of participants in the group) and % new abnormals if abnormal counts were noted. Abnormality is assessed according to standards for age and sex measurements under Quest Diagnostics criteria.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Number; unit: participants
Arm/Group | Xanthohumol | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 14
participants
  Total Red Blood Cell Count (Week 4): number of abnormals | 1 | 1
  Total Red Blood Cell Count (Week 4) : number of new abnormals | 1 | 1
  Total Red Blood Cell Count (Week 8) : number of abnormal | 0 | 1
  Total Red Blood Cell Count (Week 8) : number of new abnormals | 0 | 1
  Mean Corpuscular Hemoglobin (Week 8) : number of abnormals | 1 | 0
  Mean Corpuscular Hemoglobin (Week 8) : number of new abnormals | 1 | 0
  Hemoglobin (Week 2) : number of abnormals | 0 | 2
  Hemoglobin (Week 2) : number of new abnormals | 0 | 1
  Hemoglobin (Week 4) : number of abnormals | 2 | 2
  Hemoglobin (Week 4) : number of new abnormals | 2 | 1
  Hemoglobin (Week 6) : number of abnormals | 1 | 2
  Hemoglobin (Week 6) : number of new abnormals | 1 | 1
  Hemoglobin (Week 8) : number of abnormals | 0 | 3
  Hemoglobin (Week 8) : %new abnormals | 0 | 2
  Total White Blood Cell Count (Week 2) : number of abnormals | 3 | 2
  Total White Blood Cell Count (Week 2) : number of new abnormals | 3 | 0
  Total White Blood Cell Count (Week 4) : number of abnormals | 1 | 2
  Total White Blood Cell Count (Week 4) : number of new abnormals | 1 | 0
  Total White Blood Cell Count (Week 6) : number of abnormals | 2 | 3
  Total White Blood Cell Count (Week 6) : number of new abnormals | 2 | 1
  Total White Blood Cell Count (Week 8) : number of abnormal | 1 | 1
  Total White Blood Cell Count (Week 8) : %new abnormals | 1 | 0

13. Secondary Outcome: Total Red Blood Cell Count
Description: Enumeration of total red blood cell count. Reported as mean change from baseline.
Time Frame: Baseline, 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: mean change from baseline
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
mean change from baseline
  Total Red Blood Cell Count (Week 2) | .08 (.22) | .04 (.15)
  Total Red Blood Cell Count (Week 4) | -.06 (.20) | .04 (.20)
  Total Red Blood Cell Count (Week 6) | -.04 (.16) | .07 (.23)
  Total Red Blood Cell Count (Week 8) | .00 (.23) | .08 (.24)

14. Secondary Outcome: Total White Blood Cell Count
Description: Enumeration of total white blood cell count. Results are reported as mean change from baseline at weeks 2, 4, 6, and 8.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: thousand cells per microliter (1000/uL)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
thousand cells per microliter (1000/uL)
  Total White Blood Cell Count (Week 2) | -.05 (1.00) | -.59 (1.19)
  Total White Blood Cell Count (Week 4) | -.05 (.98) | -.09 (1.82)
  Total White Blood Cell Count (Week 6) | .23 (1.17) | -.24 (1.60)
  Total White Blood Cell Count (Week 8) | .21 (.76) | -.24 (1.44)

15. Secondary Outcome: Platelet Count
Description: Enumeration of platelet count. Results are reported as mean change from baseline at weeks 2, 4, 6, and 8.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: thousand cells per microliter (1000/uL)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
thousand cells per microliter (1000/uL)
  Platelet Count (Week 2) | 3.54 (24.05) | 2.60 (26.04)
  Platelet Count (Week 4) | 3.46 (19.62) | 0.07 (19.86)
  Platelet Count (Week 6) | 14.00 (32.01) | 22.93 (41.90)
  Platelet Count (Week 8) | 10.46 (25.62) | 7.14 (20.47)

16. Secondary Outcome: Mean Corpuscular Volume
Description: Enumeration of mean corpuscular volume (MCV). Results are reported as mean change from baseline at weeks 2, 4, 6, and 8.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
femtoliter (fL)
  Mean Corpuscular Volume (Week 2) | .14 (.76) | .20 (1.21)
  Mean Corpuscular Volume (Week 4) | .61 (1.45) | -0.27 (1.54)
  Mean Corpuscular Volume (Week 6) | .04 (1.47) | -0.25 (1.56)
  Mean Corpuscular Volume (Week 8) | .04 (.80) | -0.63 (1.88)

17. Secondary Outcome: Mean Corpuscular Hemoglobin
Description: Enumeration of mean corpuscular hemoglobin (MCH). Results are reported as mean change from baseline at weeks 2, 4, 6, and 8.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
picograms (pg)
  Mean Corpuscular Hemoglobin (Week 2) | 0.05 (0.35) | -0.06 (0.45)
  Mean Corpuscular Hemoglobin (Week 4) | 0.26 (0.53) | -0.04 (0.51)
  Mean Corpuscular Hemoglobin (Week 6) | 0.29 (0.42) | -0.13 (0.76)
  Mean Corpuscular Hemoglobin (Week 8) | 0.20 (0.52) | -0.23 (0.87)

18. Secondary Outcome: Hematocrit
Description: Enumeration of hematocrit. Results are reported as mean change from baseline at weeks 2, 4, 6, and 8.
Time Frame: 2 weeks, 4 weeks, 6 weeks, and 8 weeks.
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Placebo Oral Capsule | Xanthohumol
Number analyzed (Participants) | 14 | 16
percent (%)
  Hematocrit (Week 2) | 0.77 (1.92) | 0.48 (1.49)
  Hematocrit (Week 4) | -0.20 (1.56) | 0.23 (2.18)
  Hematocrit (Week 6) | -0.32 (1.60) | 0.57 (2.11)
  Hematocrit (Week 8) | -0.03 (2.16) | 0.44 (2.27)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Mild/Grade 1: No intervention; asymptomatic lab or radiographic findings; marginal clinical significance Moderate/Grade 2: OTC or single-physician visit; AE limited activities of daily living for <48hrs Severe/Grade 3: AE significantly limited basic self-care but did not require initial hospitalization or prolongation of hospitalization; Not immediately life-threatening but disabling Serious/Grade 4: Life threatening Serious/Grade 5: Death
Arm/Group | Xanthohumol | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 14/16 | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xanthohumol (N=16) | Placebo Oral Capsule (N=14)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (4)
Allergy symptoms (General disorders) | 3 (4) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry eyes and periorbital twitching (Eye disorders) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Indigestion (Gastrointestinal disorders) | 2 (3) | 3 (4)
Increased thirst (General disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Headache (General disorders) | 4 (4) | 3 (3)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2)
Lethargy (General disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 0 (0) | 4 (6)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hyperactivity (General disorders) | 0 (0) | 1 (1)
Shortness of breath on exertion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral edema/swelling (Vascular disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Itchy/dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Dizziness (General disorders) | 1 (1) | 0 (0)
Sore throat (General disorders) | 1 (1) | 3 (4)
Decreased urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
General body pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03735420/Prot_SAP_001.pdf